CLINICAL TRIAL: NCT05138991
Title: Assessment of the Reproducibility and Accuracy of a Portable System for Early Detection of Cardiac Dysfunction in Childhood Cancer Survivors
Brief Title: Reproducibility and Accuracy of a Portable System for Early Detection of Cardiac Dysfunction in Childhood Cancer Survivors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 21466; NCI-2021-11335 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21466 (Other: City of Hope Medical Center); P30CA033572 (NIH); R21CA261797 (NIH)
Record Dates: First submitted 2021-11-22; First posted 2021-12-01 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Screening (echo, CMR, Tonometry-based system) (Experimental): Patients undergo a one time assessment of cardiac function by echo, CMR, and the Tonometry-based system system in the clinic over 4-6 hours, and will be asked to perform their home-based measurements within 1-5 days of the clinical assessment, allowing us to directly compare measurements obtained by survivors to those by research personnel. Patients also complete questionnaires at baseline.
  Interventions: Procedure: Echocardiogram Recording; Other: Questionnaire Administration; Procedure: Stress Cardiac Magnetic Resonance Imaging; Device: Wireless Synchronized Cardiac Function Monitoring Device

INTERVENTIONS:
Procedure: Echocardiogram Recording — Undergo assessment via echo
  Other Names: Echocardiogram
Other: Questionnaire Administration — Ancillary Studies
Procedure: Stress Cardiac Magnetic Resonance Imaging — Undergo assessment via CMR
Device: Wireless Synchronized Cardiac Function Monitoring Device — SphygmoCor® Xcel Oscar 2™ Ambulatory Blood Pressure Monitor

SUMMARY:
The clinical trial compares the reproducibility and accuracy of cardiac tonometry-based portable systems that may detect early cardiac dysfunction (SphygmoCor® Xcel and Oscar 2™ ambulatory blood pressure monitor) at home and in the clinic to currently available screening tests for heart failure including echocardiogram (echo) and cardiovascular magnetic resonance (CMR). The SphygmoCor® Xcel and Oscar 2™ systems may help detect cardiac dysfunction earlier than other available screening tests because it can be self-administered outside of the clinic. This study aims to test the accuracy and practicality of these devices in the clinic setting and at home.

DETAILED DESCRIPTION:
Primary Objective(s)

Validate the accuracy of ejection fraction, as measured using a tonometry-based system (SphygmoCor® Xcel), in the clinic setting, and determine the reproducibility (Oscar 2™) at home.

Secondary Objective(s)

Determine the cost-effectiveness of tonometry-based screening in the clinic setting and at home.

ELIGIBILITY:
Inclusion Criteria:

* Previously enrolled in IRB# 14154.
* Able to understand and sign the study specific informed consent form (ICF).

Exclusion Criteria:

* Participants cannot be actively receiving cancer-directed therapy.
* Standard exclusion criteria for CMR imaging will be incorporated, and these include: implanted pacemaker or defibrillator, insulin pump, cochlear implant, central nervous system aneurismal clips, implanted neural stimulator, ocular foreign body (metal), other implanted medical devices (e.g.: drug infusion ports).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2026-07-16 (Estimated); Study Completion 2026-07-16 (Estimated)

PRIMARY OUTCOMES:
Accuracy of ejection fraction (EF) in the clinic setting, and determine its reproducibility at home. | Up to 2 years
  Validate the accuracy of ejection fraction, as measured using a tonometry-based system (SphygmoCor® Xcel), in the clinic setting, and determine the reproducibility (Oscar 2™) at home.

SECONDARY OUTCOMES:
Cost-effectiveness of tonometry-based screening in the clinic setting and at home. | Up to 2 years
  Will apply the sensitivity and specificity of echo, CMR, and the Oscar 2™ ABPM system (clinic, home-based) to compare the number of asymptomatic cardiac dysfunction cases identified via each method. Screening costs for echo and CMR, including costs of clinical services, will be obtained from the 2020 Centers for Medicare & Medicaid Services (CMS).

CONTACTS AND LOCATIONS:
Overall Officials: Saro H Armenian, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/91/NCT05138991/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-22): https://cdn.clinicaltrials.gov/large-docs/91/NCT05138991/ICF_001.pdf